CLINICAL TRIAL: NCT02043626
Title: School Wellness Policy: RCT to Implement & Evaluate Impact on Childhood Obesity
Brief Title: Study to Evaluate the Health and Wellness Policies of the New Haven Public School District.
Acronym: H&A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1008007295; 5R01HD070740 (NIH)
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Chronic Diseases; Obesity
Keywords: childhood nutrition; physical activity; school wellness; school health; nutritional policies; childhood obesity
MeSH Terms: conditions — Chronic Disease; Obesity; Motor Activity; Pediatric Obesity | interventions — Health Promotion; Marketing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physical Activity Only (Experimental): Students in 3 designated study schools will receive educational intervention and increased opportunities for physical activity.
  Interventions: Other: OPPORTUNITIES FOR PHYSICAL ACTIVITY
- Delayed Interventions Only (No Intervention): Students in 3 designated schools will receive educational interventions on health topics not related to nutrition or physical activity (i.e. peer relations, sleep, dental care, etc.)
- Nutrition and Physical Activity (Experimental): Students in 3 designated schools will receive nutrition education, nutrition standards for foods sold, and opportunities for physical activity.
  Interventions: Other: DISTRICT WELLNESS COMMITTEE; Other: NUTRITIONAL QUALITY OF FOODS AND BEVERAGES ON CAMPUS; Other: HEALTH PROMOTION AND MARKETING; Other: OPPORTUNITIES FOR PHYSICAL ACTIVITY
- Nutrition Only Interventions (Experimental): Students in 3 designated study schools will receive multiple interventions regarding nutrition education and nutrition standards for foods sold.
  Interventions: Other: NUTRITIONAL QUALITY OF FOODS AND BEVERAGES ON CAMPUS

INTERVENTIONS:
Other: DISTRICT WELLNESS COMMITTEE — Three Targeted Schools (N+PA) will expand the District's school based wellness initiative, PAW-Physical Activity and Wellness. With District support, PAW schools develop School Wellness Teams (SWTs) to identify school health priorities, implement and sustain health initiatives through school campaigns, promote healthy behavior, and support wellness policies. Results from a 3-year evaluation suggest significant and sustained positive impact on school health culture, student behavior, time-on-task, and increased physical activity among students.
  Arms: Nutrition and Physical Activity
Other: NUTRITIONAL QUALITY OF FOODS AND BEVERAGES ON CAMPUS — Policy changes will focus on 6 target schools. District will expand nutrition education by integrating other opportunities to learn and practice healthy behaviors across disciplines. Farm-to-School programs will include school visits by farmers to teach students about agriculture, healthy foods and nutrition, coinciding with Farmer's Market Menu Days. Schools will receive four 45 minute nutrition workshops per year. Community educators will offer culturally appropriate, interactive nutrition workshops and cooking demonstrations. Cafeterias will receive youth friendly nutritional messaging, regular promotion of new menu foods, and a variety of monthly nutrition-focused activities. The goals are to: increase number of students who try new menu items regularly, increase acceptance of healthy foods, and improve nutrition literacy. Policy states schools will limit celebrations that involve food to no more than 1 per class/month: 6 schools will pilot alternatives to food for celebrations.
  Arms: Nutrition Only Interventions; Nutrition and Physical Activity
Other: HEALTH PROMOTION AND MARKETING — SWP addresses health promotion and marketing by limiting product marketing in schools, expanding nutrition education and broadening health communication with parents. In 3 targeted schools, we expand to include Staff Wellness Promotion. Adults in schools are trusted and influential role models for students; by increasing their positive health behaviors, students may be influenced to adopt similar behaviors. The District will work with the City's Employee Wellness Program to increase school staff participation.
  Arms: Nutrition and Physical Activity
Other: OPPORTUNITIES FOR PHYSICAL ACTIVITY — District-wide policies include mandates for daily physical activity and PE and development of policies that prohibit withholding PE for punitive reasons. To further increase physical activity, the School Wellness Policy specifies expanding programs/activities that meet need, interest, and abilities of students. Exer-gaming consoles will be provided to 6 schools and will be integrated into 5th-8th grade PE classes and after-school programs. New and innovate gym equipment will be purchased for the 6 target schools for use in gym class and after school programming. Various pedometer and interactive programs encouraging physical activity in and outside of school are planned for the 6th grade.
  Arms: Nutrition and Physical Activity; Physical Activity Only

SUMMARY:
Our long-term objective is to reduce the rates and risk of childhood obesity via school-based nutrition and physical activity policies. Using a randomized design, we propose to monitor and evaluate how Connecticut's first-ranked District Wellness Policy, in the New Haven Public School district, is implemented and determine its impact on children's obesogenic behaviors, weight outcomes, and school performance. This study is designed to significantly advance empirical research on school wellness policies and to provide important evidence to guide future interventions in schools and communities - translating science to improved health of the public.

DETAILED DESCRIPTION:
Consistent with NIH priorities, our long-term objective is to reduce the rates and risk of childhood obesity via school-based nutrition and physical activity policies. We propose to monitor and evaluate how Connecticut's first-ranked School Wellness Policy, in the New Haven Public School district, is implemented and determine its impact on children's obesogenic behaviors, weight outcomes, and school performance. We will evaluate a strategy of implementation at 12 targeted schools using a randomized design. Focusing on targeted schools will enable a more rigorous evaluation of School Wellness Policy implementation, barriers/facilitators, and ultimately the behavioral and health impacts of school-based policies on childhood obesity. We propose a multi-level assessment of factors that may influence childhood obesity using the Ecological Model as a guiding framework.

Thus we propose a multi-sectoral, multi-level approach, focused on children, families, schools, and community. This ambitious project is possible because of the expertise and strong collaborative partnerships between The New Haven Public Schools and two Yale University research centers: The Rudd Center for Food Policy and Obesity and CARE: Community Alliance for Research and Engagement. Our partnership builds on Principles and Guidelines for Community-University Research Partnerships developed by a 12-member committee of community and university leaders and endorsed by Yale University and community partners in 2009.

This study is designed to significantly advance empirical research on school wellness policies: focused on implementation and measurable impact on student health. No matter how well written, a school wellness policy must be effectively implemented to achieve its potential impact. Further, students within schools represent only two components of a larger socio-ecological system that influences eating behavior, physical activity, and weight status. The federal mandate for school wellness policies requires districts to address many aspects of the school environment (e.g., nutrition education, nutrition standards for foods sold, and opportunities for physical activity). To maximize improvements, this type of multi-component policy is needed. However, this complexity makes it difficult to evaluate policy impact and draw conclusions about the causal relationships between specific policies and student health. With our team's unique strengths and these challenges in mind, we designed this research study with the following Specific Aims:

1. Track and evaluate a strategy of targeted implementation of a School Wellness Policy.
2. Identify factors that facilitate or impede implementation of The School Wellness Policy, including neighborhood, school, and student determinants; and
3. Evaluate the impact of implementation of The School Wellness Policy on obesogenic behaviors and health outcomes as well as school performance.

We will collaborate with the District to implement a subset of nutrition and physical activity policies in 12 schools using a randomized 2 x 2 research design. This will permit comparison of the potential unique and synergistic effects of these nutrition and physical activity policies on student behaviors and related health outcomes. We will follow a cohort of 5th grade students (N≈700) annually for four years to assess potential changes to student eating behaviors, physical activity levels, and BMI. We use a multi-method approach to collect data and examine predictors of these outcomes from across levels of the socio-ecological framework: student variables, family characteristics, school policies, and neighborhood features.

This multidisciplinary proposal is synchronous with specific research objectives articulated in Program Announcement (PA-10-052) School Nutrition and Physical Activity Policies, Obesogenic Behaviors and Weight Outcomes. As noted, few studies to date have examined the policy implementation process. We directly target the implementation and impact of health-related policies in schools, measuring obesogenic behaviors and BMI as primary outcomes. We have an active tracking system to monitor impact of policies, and we focus on minority populations traditionally vulnerable and underserved. As stated by NIH in this program announcement, policy-based approaches to combat obesity in schools exist; however, knowledge is lacking in key areas concerning the optimal policies, key implementation strategies for such policies, and the impact of these policies on important health and social outcomes. The proposed project will advance scientific knowledge and understanding in this arena and provide important evidence to guide future interventions in schools and communities translating science to improved health of the public.

ELIGIBILITY:
Inclusion Criteria:

* Student of the New Haven School District--State of Connecticut
* Enrolled in 12 eligible schools participating in study
* Child between the ages of 9 and 14 or in grades 5-8 as of the fall of 2011
* Primary Language of communication is English

Exclusion Criteria:

* Not enrolled in one of 12 participating schools
* Not in target grade (5-8) as of the fall 2011

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 796 (Actual)
Dates: Start 2011-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI). | Baseline through Follow-up: Grades 5-6-7-8
  Body weight and height to calculate BMI annually from baseline (grade 5) through follow-up (grade 8)

SECONDARY OUTCOMES:
Change in student nutritional habits (eating behaviors). | Baseline through Follow-up: Grades 5-6-7-8
  Surveying student nutritional habits and close observation of nutritional habits (food consumed) in school.
Change in level of physical activity. | Baseline through Follow-up: Grades 5-6-7-8
  Surveying of student physical activity habits and observation of student participation in class time or after school physical activity programs.
Mental Health | Baseline through Follow-up: Grades 5-6-7-8
  Strengths and Difficulties Questionnaire screens child mental health problems, five subscales: emotional problems, hyperactivity, relationship, conduct and pro-social behavior.
Standardized test scores | Baseline through Follow-up: Grades 5-6-7-8
  Standardized test scores, reading and mathematics

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Ickovics, PHD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Ickovics JR, Carroll-Scott A, Peters SM, Schwartz M, Gilstad-Hayden K, McCaslin C. Health and academic achievement: cumulative effects of health assets on standardized test scores among urban youth in the United States. J Sch Health. 2014 Jan;84(1):40-8. doi: 10.1111/josh.12117. PMID 24320151
- [Background] Kallem S, Carroll-Scott A, Rosenthal L, Chen E, Peters SM, McCaslin C, Ickovics JR. Shift-and-persist: a protective factor for elevated BMI among low-socioeconomic-status children. Obesity (Silver Spring). 2013 Sep;21(9):1759-63. doi: 10.1002/oby.20195. Epub 2013 May 13. PMID 23671041
- [Background] Kallem S, Carroll-Scott A, Gilstad-Hayden K, Peters SM, McCaslin C, Ickovics JR. Children's report of lifestyle counseling differs by BMI status. Child Obes. 2013 Jun;9(3):216-22. doi: 10.1089/chi.2012.0100. Epub 2013 Apr 30. PMID 23631343
- [Background] Wang S, Schwartz MB, Shebl FM, Read M, Henderson KE, Ickovics JR. School breakfast and body mass index: a longitudinal observational study of middle school students. Pediatr Obes. 2017 Jun;12(3):213-220. doi: 10.1111/ijpo.12127. Epub 2016 Mar 17. PMID 26989876
- [Background] Carroll-Scott A, Gilstad-Hayden K, Rosenthal L, Eldahan A, McCaslin C, Peters SM, Ickovics JR. Associations of Neighborhood and School Socioeconomic and Social Contexts With Body Mass Index Among Urban Preadolescent Students. Am J Public Health. 2015 Dec;105(12):2496-502. doi: 10.2105/AJPH.2015.302882. Epub 2015 Oct 15. PMID 26469652
- [Background] Chandler I, Rosenthal L, Carroll-Scott A, Peters SM, McCaslin C, Ickovics JR. Adolescents Who Visit the Emergency Department Are More Likely to Make Unhealthy Dietary Choices: An Opportunity for Behavioral Intervention. J Health Care Poor Underserved. 2015 Aug;26(3):701-11. doi: 10.1353/hpu.2015.0086. PMID 26320906
- [Background] Schwartz DL, Gilstad-Hayden K, Carroll-Scott A, Grilo SA, McCaslin C, Schwartz M, Ickovics JR. Energy drinks and youth self-reported hyperactivity/inattention symptoms. Acad Pediatr. 2015 May-Jun;15(3):297-304. doi: 10.1016/j.acap.2014.11.006. Epub 2015 Feb 9. PMID 25676784
- [Background] Schwartz MB, Gilstad-Hayden K, Henderson KE, Luedicke J, Carroll-Scott A, Peters SM, McCaslin C, Ickovics JR. The Relationship between Parental Behaviors and Children's Sugary Drink Consumption Is Moderated by a Television in the Child's Bedroom. Child Obes. 2015 Oct;11(5):560-8. doi: 10.1089/chi.2014.0041. Epub 2015 Aug 28. PMID 26317365
- [Background] Rosenthal L, Earnshaw VA, Carroll-Scott A, Henderson KE, Peters SM, McCaslin C, Ickovics JR. Weight- and race-based bullying: health associations among urban adolescents. J Health Psychol. 2015 Apr;20(4):401-12. doi: 10.1177/1359105313502567. Epub 2013 Oct 22. PMID 24155192
- [Background] Jernigan MM, Rosenthal L, Carroll-Scott A, Peters SM, McCaslin C, Ickovics JR. Emotional Health Predicts Changes in Body Mass Index (BMI-z) Among Black and Latino Youth. Clin Pediatr (Phila). 2015 Jun;54(7):693-6. doi: 10.1177/0009922815574080. Epub 2015 Feb 26. No abstract available. PMID 25724990
- [Background] Smith LP, Gilstad-Hayden K, Carroll-Scott A, Ickovics J. High waist circumference is associated with elevated blood pressure in non-Hispanic White but not Hispanic children in a cohort of pre-adolescent children. Pediatr Obes. 2014 Dec;9(6):e145-8. doi: 10.1111/ijpo.246. Epub 2014 Jul 3. PMID 24990227
- [Background] Gilstad-Hayden K, Carroll-Scott A, Rosenthal L, Peters SM, McCaslin C, Ickovics JR. Positive school climate is associated with lower body mass index percentile among urban preadolescents. J Sch Health. 2014 Aug;84(8):502-6. doi: 10.1111/josh.12177. PMID 25040118
- [Background] Earnshaw VA, Rosenthal L, Carroll-Scott A, Peters SM, McCaslin C, Ickovics JR. Teacher Involvement as a Protective Factor from the Association between Race-Based Bullying and Smoking Initiation. Soc Psychol Educ. 2014 Jun 1;17(2):197-209. doi: 10.1007/s11218-014-9250-1. PMID 24955021
- [Background] Carroll-Scott A, Gilstad-Hayden K, Rosenthal L, Peters SM, McCaslin C, Joyce R, Ickovics JR. Disentangling neighborhood contextual associations with child body mass index, diet, and physical activity: the role of built, socioeconomic, and social environments. Soc Sci Med. 2013 Oct;95:106-14. doi: 10.1016/j.socscimed.2013.04.003. Epub 2013 Apr 10. PMID 23642646
- [Derived] Ickovics JR, Duffany KO, Shebl FM, Peters SM, Read MA, Gilstad-Hayden KR, Schwartz MB. Implementing School-Based Policies to Prevent Obesity: Cluster Randomized Trial. Am J Prev Med. 2019 Jan;56(1):e1-e11. doi: 10.1016/j.amepre.2018.08.026. PMID 30573151
- [Derived] Assoumou SA, Wang J, Tasillo A, Eftekhari Yazdi G, Tsui JI, Strick L, Linas BP. Hepatitis C Testing and Patient Characteristics in Washington State's Prisons Between 2012 and 2016. Am J Prev Med. 2019 Jan;56(1):8-16. doi: 10.1016/j.amepre.2018.08.016. Epub 2018 Nov 19. PMID 30467088